CLINICAL TRIAL: NCT01108848
Title: Patient Registry for Berinert®, a C1-Esterase Inhibitor
Brief Title: Patient Registry Study of Berinert® in Normal Clinical Practice
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CE1145_5002; 1500 (Other: CSL Behring)
Record Dates: First submitted 2010-04-12; First posted 2010-04-22 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Includes: Hereditary Angioedema
Keywords: C1-esterase Inhibitor; Hereditary angioedema; Acute HAE attack
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Berinert: Patients requiring treatment with Berinert®
  Interventions: Biological: Berinert® (C1 Esterase Inhibitor)

INTERVENTIONS:
Biological: Berinert® (C1 Esterase Inhibitor) — Berinert® is marketed as a lyophilized concentrate available in a single-use vial to be reconstituted with sterile water before administration as described in the prescribing information.
  Other Names: C1-INH; Berinert P; CE1145

SUMMARY:
The objective of this patient registry is to collect data on the safety of Berinert® in normal clinical practice in the United States. The patient registry will be maintained for a period of at least 3 years. The duration of individual patient participation will vary and is determined by the frequency of hereditary angioedema (HAE) attacks and the patient's need for Berinert® treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any patient receiving CSL Behring's C1-esterase inhibitor
* Written informed consent (may not be required for some retrospective chart review cases)

Exclusion Criteria:

* Any patient participating in an HAE study using other C1-inhibitors than Berinert®

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An attempt will be made to prospectively identify patients and enroll them into this registry before treatment is required. In addition, retrospective chart/case review and data collection may be conducted.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of thrombotic and thrombo-embolic events | Within 30 days of treatment with Berinert®
Occurrence of suspected viral transmission | Duration of the study, at least 3 years
Use of concomitant medications and plasma products | Duration of the study, at least 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Program Director, Study Director — CSL Behring
Locations (40):
- United States (34):
  - United States, Arizona, Scottsdale, Arizona
  - United States, California, Granada Hills, California
  - United States, California, Los Angeles, California
  - United States, California, Redding, California
  - United States, California, San Diego, California
  - United States, Georgia, Atlanta, Georgia
  - United States, Idaho, Idaho Falls, Idaho
  - United States, Louisiana, New Orleans, Louisiana
  - United States, Maryland, Chevy Chase, Maryland
  - United States, Maryland, Columbia, Maryland
  - United States, Massachusetts, Boston, Massachusetts
  - United States, Minnesota, Plymouth, Minnesota
  - United States, Missouri, Kansas City, Missouri
  - United States, Missouri, St Louis, Missouri
  - United States, New Jersey, Branchburg, New Jersey
  - United States, New Jersey, Edison, New Jersey
  - United States, New Jersey, Iselin, New Jersey
  - United States, New Jersey, Ocean City, New Jersey
  - United States, New York, New York, New York
  - United States, New York, North Syracuse, New York
  - United States, North Carolina, Durham, North Carolina
  - United States, Ohio, Centerville, Ohio
  - United States, Ohio, Cincinnati, Ohio
  - United States, Oklahoma, Oklahoma City, Oklahoma
  - United States, Oklahoma, Tulsa, Oklahoma
  - United States, Oregon, Lake Oswego, Oregon
  - United States, Pennsylvania, Altoona, Pennsylvania
  - United States, Pennsylvania, Hershey, Pennsylvania
  - United States, Pennsylvania, Pittsburgh, Pennsylvania
  - United States, South Carolina, Columbia, South Carolina
  - United States, South Dakota, Rapid City, South Dakota
  - United States, Texas, Dallas, Texas
  - United States, Washington, Spokane, Washington
  - United States, Washington, Tacoma, Washington
- Denmark, Odense C, Odense C, Denmark
- Germany (4):
  - Germany, Mainz, Mainz, Germany
  - Germany, Berlin, Berlin
  - Germany, Frankfurt, Frankfurt
  - Germany, München, München
- Switzerland, Luzern 16, Lucerne, Switzerland

REFERENCES:
- [Derived] Bygum A, Martinez-Saguer I, Bas M, Rosch J, Edelman J, Rojavin M, Williams-Herman D; Berinert Registry Investigators. Use of a C1 Inhibitor Concentrate in Adults >/=65 Years of Age with Hereditary Angioedema: Findings from the International Berinert(R) (C1-INH) Registry. Drugs Aging. 2016 Nov;33(11):819-827. doi: 10.1007/s40266-016-0403-0. PMID 27699634
- [Derived] Busse P, Bygum A, Edelman J, Lumry W, Machnig T, Martinez-Saguer I, Rojavin M. Safety of C1-esterase inhibitor in acute and prophylactic therapy of hereditary angioedema: findings from the ongoing international Berinert patient registry. J Allergy Clin Immunol Pract. 2015 Mar-Apr;3(2):213-9. doi: 10.1016/j.jaip.2014.08.014. Epub 2014 Oct 29. PMID 25609333
- See also: Hereditary Angioedema Association (HAEA) — http://www.hereditaryangioedema.com/